CLINICAL TRIAL: NCT07389174
Title: An Open-Label, Exploratory Study to Evaluate the Safety and Preliminary Efficacy of LC-K76 in Combination With Endocrine Therapy in Patients With Metastatic Hormone-Sensitive Prostate Cancer
Brief Title: Safety and Efficacy Evaluation of LC-K76 in Patients With Metastatic Hormone-Sensitive Prostate Cancer
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Ren Shancheng, Professor, Chief of Urology, Shanghai Changzheng Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LC-K76-101
Record Dates: First submitted 2025-12-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: mHSPC; mHNPC; Prostate Cancer Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High-Volume mHSPC: Standard of Care (Active Comparator): Participants with high-volume metastatic hormone-sensitive prostate cancer (mHSPC). Participants in this arm receive standard-of-care endocrine therapy alone.
  Interventions: Drug: Standard Endocrine Therapy
- High-Volume mHSPC: LC-K76 + Standard Endocrine Therapy (Experimental): Participants with high-volume metastatic hormone-sensitive prostate cancer (mHSPC). High volume is defined as the presence of visceral metastases or ≥ 4 bone lesions with ≥ 1 beyond the vertebral bodies and pelvis. Participants in this arm receive oral LC-K76 combined with standard-of-care endocrine therapy.
  Interventions: Drug: Standard Endocrine Therapy; Dietary Supplement: LC-K76
- Low-Volume mHSPC: LC-K76 + Standard Endocrine Therapy (Experimental): Participants with low-volume metastatic hormone-sensitive prostate cancer (mHSPC). Low volume is defined as ≤ 3 bone metastases confined to the vertebral bodies and pelvis, and no visceral metastases. Participants in this arm receive oral LC-K76 combined with standard-of-care endocrine therapy.
  Interventions: Drug: Standard Endocrine Therapy; Dietary Supplement: LC-K76
- Low-Volume mHSPC: Standard of Care (Active Comparator): Participants with low-volume metastatic hormone-sensitive prostate cancer (mHSPC). Participants in this arm receive standard-of-care endocrine therapy alone.
  Interventions: Drug: Standard Endocrine Therapy

INTERVENTIONS:
Drug: Standard Endocrine Therapy — Participants in this arm receive the standard-of-care endocrine therapy for metastatic hormone-sensitive prostate cancer (mHSPC). This regimen consists of Androgen Deprivation Therapy (ADT) (e.g., Goserelin, Leuprorelin, Triptorelin, or Degarelix) combined with an oral Androgen Receptor (AR) inhibitor (e.g., Apalutamide, Enzalutamide, Darolutamide, Rezvilutamide, or Abiraterone Acetate). The specific choice of drugs is determined by the investigator based on approved clinical use .
Dietary Supplement: LC-K76 — Oral administration at a dose of 1.2 g twice daily (BID), taken 30 minutes before breakfast and dinner, for a treatment period of 24 weeks.
  Arms: High-Volume mHSPC: LC-K76 + Standard Endocrine Therapy; Low-Volume mHSPC: LC-K76 + Standard Endocrine Therapy

SUMMARY:
This study is a single-centre, randomised, paired 24-week intervention dosing trial. Its purpose is to evaluate the safety profile and efficacy of the investigational drug in subjects with metastatic hormone-sensitive prostate cancer receiving oral LC-K76 treatment.

Following a screening period not exceeding three weeks, subjects will enter a one- to two-week matching and randomization phase. Subsequently, subjects will be assigned to receive the study drug for a 24-week treatment period, followed by a 24-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Male, aged ≥ 18 years.
2. Histologically or cytologically confirmed newly diagnosed metastatic hormone-sensitive prostate adenocarcinoma, without small cell carcinoma or small cell components.
3. Presence of at least one bone metastasis or visceral metastasis (excluding lymph nodes) detected by systemic imaging (CT/MRI).
4. No prior treatment for prostate cancer before enrollment (including but not limited to radical surgery, radiotherapy, endocrine therapy, or chemotherapy).
5. No history of allergy to dandelion or dandelion products.
6. ECOG performance status ≤ 2.
7. Plan to receive and maintain Androgen Deprivation Therapy (ADT) combined with an androgen receptor antagonist (e.g., enzalutamide, apalutamide, darolutamide), abiraterone acetate, or other drugs inhibiting testosterone synthesis during the study period.
8. Subjects are able to comply with oral LC-K76 capsule administration and adhere to study requirements throughout the study

Exclusion Criteria:

1. Lack of pathological evidence for prostate cancer diagnosis.
2. Prior receipt of any treatment modality for prostate cancer.
3. Patients with other primary malignant tumors that were progressive or required active treatment within the past 3 years.
4. Patients with diabetes requiring continuous insulin therapy or poorly controlled diabetes.
5. Known or suspected central nervous system metastases or active leptomeningeal disease.
6. Significant abnormalities in bone marrow, coagulation, renal, and hepatic function, defined as laboratory values at randomization: Hemoglobin < 90 g/L, Neutrophils < 1.5 × 10$^9$/L, Platelets < 75 × 10$^9$/L, ALT > 2.5 × ULN, AST > 2.5 × ULN, or Serum Total Bilirubin > 1.5 × ULN; eGFR < 60 mL/min/1.73m$^2$.
7. Any severe disease affecting cardiopulmonary function or high-risk conditions.
8. History of severe drug allergies.
9. Presence of factors interfering with swallowing, chronic diarrhea, intestinal obstruction, or other factors affecting drug intake and absorption.
10. Concurrent psychiatric illness or neurological symptoms judged to make participation difficult.
11. Any condition that, in the judgment of the investigator, poses a severe safety risk to the patient, may confound study results, or may affect the patient's ability to complete the study (e.g., poorly controlled hypertension, severe diabetes, neurological or psychiatric disorders), or any other relevant conditions.
12. Concurrent participation in other clinical trials or use of other investigational drugs.
13. Refusal or inability to sign the informed consent form.

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | From baseline to primary completion, which may take up to 24 to 48 weeks
  The Incidence of Adverse Events is defined as the proportion of subjects in a clinical trial who experience at least one Adverse Event (AE) during the defined observation period, which is assessed by CTCAE 5.0.

SECONDARY OUTCOMES:
PSA Undetectable Rate | From baseline to primary completion, which may take up to 24 to 48 weeks
  Percentage of participants who convert from detectable PSA (≥ 0.2 ng/mL) at baseline to undetectable PSA (< 0.2 ng/mL) during the study.
PSA Response Rate | From baseline to primary completion, which may take up to 24 to 48 weeks
Time to CRPC（Castration-Resistant Prostate Cancer） | From baseline to primary completion, which may take up to 24 to 48 weeks
Disease Control Rate (DCR) | From baseline to primary completion, which may take up to 24 to 48 weeks
  Defined as the proportion of subjects whose best overall response, assessed per standardized criteria (RECIST 1.1 and PCWG3), is Complete Response (CR), Partial Response (PR), or Stable Disease (SD) .
Radiographic Progression-Free Survival （rPFS ） | From baseline to primary completion, which may take up to 24 to 48 weeks
  Defined as the time from randomization to the first objective evidence of disease progression as assessed by radiographic imaging, or death from any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (1):
- Changzheng hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No